CLINICAL TRIAL: NCT03123874
Title: Milk in Life Conditions (MiLC): Characterizing the Bacterial Composition of Human Milk Pumped and Stored in "Real-life" Conditions
Brief Title: Milk in Life Conditions (MiLC): Bacterial Composition of Human Milk Pumped and Stored in "Real-Life" Conditions
Acronym: MiLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Idaho (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #: 1608006566; 2T32DK007158-42 (NIH); NYC-399436 (Other Grant/Funding Number: NIFA/USDA)
Record Dates: First submitted 2017-04-06; First posted 2017-04-21 (Actual); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-04

CONDITIONS: Human Milk Microbiome; Bacterial Growth
Keywords: human milk; breast milk; expressed human milk; bacterial communities; microbiome; breast pump; bacterial growth
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: All participants will pump their milk with two pump set-ups: own and sterile supplies. The pump set-up each woman used first was randomized according to infant feeding status (human milk only vs. human milk and complementary foods).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sterile pump set-up first (Experimental): Participants will pump with sterile pump set-ups first. Approximately 3 hours later, participants will pump with their own pump set-ups.
  Interventions: Device: Sterile pump set-up; Device: Mother's Own pump set-up
- Mother's Own pump set-up first (Experimental): Participants will pump with their own pump set-ups first. Approximately 3 hours later, participants will pump with sterile pump set-ups.
  Interventions: Device: Sterile pump set-up; Device: Mother's Own pump set-up

INTERVENTIONS:
Device: Sterile pump set-up — Medela symphony breast pump (model number 0240108) and disposable, sterile collection kits (model number 67399S).
Device: Mother's Own pump set-up — Mother's own electric breast pump and own collection kit (previously used and cleaned at home using her usual practices).

SUMMARY:
The MiLC trial is a randomized control trial of two different breast pump set-ups: mother's own and sterile. The objective of this trial is to investigate the bacterial composition of human milk pumped and stored in "real-life" conditions. To meet this objective, lactating mothers will fully express breast milk from one breast on two consecutive pumping sessions at home, once with the participant's own pumps and collection kits (own pump set-up) and once with a hospital-grade pump and disposable, sterile collection kits (sterile pump set-up). Randomization will be used to determine which pump participants use first. From the total volume of milk pumped during each pumping session, the researchers will collect 1 oz. Milk from both pumps will be stored at home and sampled on days 0, 2, 4, and 30 after expression for analysis of its bacterial composition.

DETAILED DESCRIPTION:
Participants will donate 1 oz of human milk during each of two consecutive pumping sessions, for a total volume of 2 oz donated on one day. To collect this human milk, participants will be asked to fully express one breast during each pumping session. Participants will pump once with the participant's own pump set-up and once with the sterile pump set-up (provided by the research team). Women will be randomized to which pump is used first.

Randomization will be done using stratified randomization as follows: participants were stratified by how their infants were fed, namely whether infants were fed human milk only vs. human milk and complementary foods). Then, randomization was conducted within each strata. The researchers aim to have a minimum of 25 participants in each stratum.

All human milk collections will occur at participants' homes between 0700 and 1100 hours. The second pumping session must begin 3 hours (+/-30 minutes) after the beginning of the first pumping session (e.g. the first pumping session at 7:30 am and the second at 10:30 am). Participants will elect from which breast to donate human milk and that breast will be used for both pumping sessions. Participants will be asked not to nurse from or pump that breast during the 2 hours before the first pumping session and not until after the second pumping session (a total of ~5.5 hours).

From the milk produced during each pumping session (which could be up to ~6 oz), researchers will collect 1 oz using a sterile, plastic syringe. Participants will keep the remaining volume of milk. Each ounce of milk collected will be separated into 5 sterile containers (provided). Participants will store donated milk at home until it is picked up by a researcher 2, 4, and 30 days after pumping.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women over the age of 18 years
* Self-reported as healthy women and infants
* Use an electric breast pump
* Confident of ability to donate 1 oz of milk from one breast during each of two consecutive pumping sessions where pumping sessions are 3 hours (+/- 30 minutes) apart and between 0700-1100 hours.
* Able to store donated milk at home for 30 days
* Have infants who do not consume formula or only consume formula episodically as long as the most recent formula-feeding occurred > 2 weeks before the day milk is pumped for this study.

Exclusion Criteria:

* Not confident of ability to donate 1 oz of milk from one breast during each of two consecutive pumping sessions, 3 hours (+/- 30 minutes) apart and between the hours of 0700-1100 hours.
* Infant consumption of formula in the past 2 weeks
* Current indication of breast infection (e.g., breast pain, discomfort, lumps, mastitis with fever, red streaks, or hard red portions of the breast)
* Breast pain that the woman does not consider "normal" for lactation/breastfeeding
* Signs/symptoms of acute illness in woman or infant in past 7 days including fever (rectal or temporal temperature ≥99.5 F), dark green nasal discharge, diarrhea (abrupt onset of 3 or more excessively "loose" stools in one day), vomiting (where infant vomiting is not associated with feeding), or severe cough.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M. Rasmussen, ScD, Principal Investigator — Cornell University; Anthony Hay, PhD, Principal Investigator — Cornell University; Sarah Reyes, MS, Study Director — Cornell University
Locations (1):
- Hay Laboratory, B75C Wing Hall, Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers are currently undecided about how all the data from the study will be released but 16S rRNA data will be released through INSDC (the International Nucleotide Sequence Database Collaboration, which encompasses NCBI, EBI and DDBJ).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sterile Pump Set-up First | Mother's Own Pump Set-up First
Started | 27 | 25
Completed | 27 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sterile Pump Set-up First | Mother's Own Pump Set-up First | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (4.1) | 33.6 (4.0) | 33.6 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/white | 23 | 22 | 45
  African American/black | 0 | 1 | 1
  Asian or Pacific Islander | 2 | 1 | 3
  Native American | 1 | 0 | 1
  Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52
Infant feeding status, number fed human milk only [Count of Participants; unit: Participants] | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Community Richness
Description: Richness is the total number of different bacterial taxa detected in the sample. This metric will be assessed on data collected via high-throughput sequencing of the bacterial 16S rRNA gene present in milk.
Time Frame: 0 days after pumping
Population: Data analyzed for all participants
Measure: Mean (Standard Deviation); unit: Observed taxa
Arm/Group | Sterile Pump Set-up First | Mother's Own Pump Set-up First
Number analyzed (Participants) | 27 | 25
Observed taxa
  In Milk Collected with Sterile Pump Set-Up | 64.2 (38.3) | 58.9 (26.9)
  In Milk Collected with Mother's Own Pump Set-Up | 64.0 (30.7) | 60.8 (32.8)
Statistical Analysis 1: Comparison: Sterile Pump Set-up First vs Mother's Own Pump Set-up First; Test type: Other — Linear mixed effects models testing the effect of pump set-up on the number of live aerobic bacterial counts. The fixed effect of interest will be pump set-up. Model will also be adjusted for infant feeding status (human milk only vs. human milk and complementary foods) and randomization schedule (which pump set-up went first); p = 0.9, Mixed Models Analysis — Results were considered statistically significant at p<0.05. No adjustments were made to p-values; Mean Difference (Final Values) = 0.827 — Ratio of mean bacterial taxa in milk collected with own / sterile pump set-ups

2. Primary Outcome: Bacterial Community Diversity
Description: Bacterial community diversity will be assessed using the the Shannon diversity index. The Shannon diversity index is a type of entropy measure and is a function of the distribution of the total number of organisms across all of the species. If S is the total number of species in the sample and p_i is the number of organisms in the i-th species divided by the total number of organisms, then Diversity = -Σ p_i log(p_i). This metric will be assessed on data collected via high-throughput sequencing of the bacterial 16S rRNA gene present in milk.
Time Frame: 0 days after pumping
Population: Data analyzed from all participants.
Measure: Mean (Standard Deviation); unit: Shannon Diversity Index
Arm/Group | Sterile Pump Set-up First | Mother's Own Pump Set-up First
Number analyzed (Participants) | 27 | 25
Shannon Diversity Index
  In Milk Collected with Sterile Pump Set-Up | 3.89 (1.18) | 3.56 (1.13)
  In Milk Collected with Mother's Own Pump Set-Up | 3.84 (1.08) | 3.93 (1.26)
Statistical Analysis 1: Comparison: Sterile Pump Set-up First vs Mother's Own Pump Set-up First; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3, Mixed Models Analysis — Results were considered statistically significant at p<0.05. No adjustments were made to p-values; Mean Difference (Final Values) = 0.163 — Ratio of mean Shannon Diversity Index in milk collected with own / sterile pump set-ups

3. Primary Outcome: Total Live Aerobic Bacterial Counts
Description: Number of live total aerobic bacteria in milk assessed by aerobic culturing of milk on plate count agar. Reported as colony-forming units (CFU)/mL.
Time Frame: 0 days after pumping
Population: Data for all participants analyzed.
Measure: Geometric Mean (Standard Deviation); unit: Colony-forming units (CFU)/mL
Groups:
- Sterile Pump Set-up First: Participants will pump with sterile pump set-ups first. Approximately 3 hours later, participants will pump with their own pump set-ups.
  Sterile pump set-up: Medela symphony breast pump (model number 0240108) and disposable, sterile collection kits (model number 67399S).
  Mom's own pump set-up: Mom's own electric breast pump and own collection kit (previously used and cleaned at home using her usual practices).
- Own Pump Set-up First: Participants will pump with their own pump set-ups first. Approximately 3 hours later, participants will pump with sterile pump set-ups.
  Sterile pump set-up: Medela symphony breast pump (model number 0240108) and disposable, sterile collection kits (model number 67399S).
  Mom's own pump set-up: Mom's own electric breast pump and own collection kit (previously used and cleaned at home using her usual practices).
Arm/Group | Sterile Pump Set-up First | Own Pump Set-up First
Number analyzed (Participants) | 27 | 25
Colony-forming units (CFU)/mL
  In Milk Collected with Sterile Pump Set-Up | 1848 (734) | 1233 (490)
  In Milk Collected with Mother's Own Pump Set-Up | 9157 (3638) | 6109 (2427)
Statistical Analysis 1: Comparison: Sterile Pump Set-up First vs Own Pump Set-up First; Test type: Other — Linear mixed effects models testing the effect of pump set-up on the number of live aerobic bacterial counts. The fixed effect of interest will be pump set-up. Model will also be adjusted for infant feeding status (human milk only vs. human milk and complementary foods) and randomization schedule (which pump set-up went first). Random effect was participant ID to account for multiple samples for each participant; p = 0.0003, Mixed Models Analysis — Results were considered statistically significant at p<0.05. No adjustments were made to p-values; Mean Difference (Final Values) = 4.95 — Ratio of mean bacterial counts in milk collected with own / sterile pump set-ups

ADVERSE EVENTS:
Time Frame: No adverse events data collected for this study
Description: No adverse events data collected for this study
Arm/Group | Sterile Pump Set-up First | Mother's Own Pump Set-up First
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03123874/Prot_SAP_000.pdf